CLINICAL TRIAL: NCT06678633
Title: Safety and Usability of the T-Control® Catheter in Cytostatics Management: a Pilot Study
Brief Title: T-Control® Safety for Cytostatics Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rethink Medical SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: RM-TCONTROL-2025-06
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Non-muscle-invasive Bladder Cancer
Keywords: Intravesical therapy; Inmunotherapy; Chemotherapy; Non-muscle-invasive bladder cancer; Foley catheter; Bladder instillation
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Comparative, randomised, prospective and crossover pilot study with two arms
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- T-Control® (Experimental): Patients will be catheterized for intravesical therapy with a new Foley-type silicone catheter with an integrated fluid-control valve into the catheter's distal end.
  Interventions: Device: T-Control® (experimental)
- Folysil® (Active Comparator): Patients will be catheterized for intravesical therapy with Folysil® Silicone catheter (Coloplast), the usual clinical practice in the participating center.
  Interventions: Device: Folysil® (control)

INTERVENTIONS:
Device: T-Control® (experimental) — Patients will receive intravesical therapy (1-2 hours) through T-Control®, a new Foley-type silicone catheter with an integrated fluid-control valve into the catheter's distal end, which has three positions.
  Arms: T-Control®
Device: Folysil® (control) — Patients will receive intravesical therapy (1-2 hours) through Folysil® Silicone catheter (Coloplast), the usual clinical practice in the participating center.
  Arms: Folysil®

SUMMARY:
The goal of this pilot clinical trial is to know if this study is feasable in terms of design, recruitment and interventions, as well as gather preliminary data to determine if the T-Control® catheter is safer than the conventional Foley-type catheter during intravesical therapy with oncological patients. It will also learn about the usability of T-Control®. The main questions it aims to answer are:

* Does T-Control® lower the rate of spillages occurred during intravesical treatments?
* Is T-Control® a better device in terms of usability during intravesical treatments?

Researchers will compare T-Control® catheter to a conventional Foley-type catheter (Folysil® Silicone catheter, Coloplast) to see if T-Control® reduce the rate of accidental spillages.

Participants will:

* Undergo intravesical therapy with the 2 devices used in the study (in two seuqencial cycles of intravesical treatment): T-Control® catheter (experimental intervention) or Folysil® silicone catheter (control intervention).
* At the end of the procedure (1-2 hours), the catheter will be removed or changed. During the first visit, patients will be catheterised with the catheter for the randomly assigned intervention, while in the subsequent visit they will be catheterised with the alternate catheter.
* Healthcare professionals involved in the procedure will take note of spillages and others adverse events occurred during the intravesical instillation.
* At the end of the study, healthcare proffesionals will evaluate the usability perceived of both devices used for intravesical treatment.

DETAILED DESCRIPTION:
This is a comparative, randomised, prospective and crossover pilot study with two arms that aims to compare the T-Control® catheter versus a conventional Foley-type catheter (Folysil®, Colopalst) in bladder cancer patients who require intravesical chemotherapy or immunotherapy treatment, monitoring the patient from the insertion of the catheter until its removal or change (1 to 2 hours) during each of the two visits programmed for the study (one for each treatment).

The general purpose of this pilot study is to determine the feasibility of a clinical study analysing the advantages that T-Control® can provide, compared with usual clinical practice in the participating center, with respect to chemotherapy and immunotherapy administration and waste management in a prospective, randomised, comparative crossover pilot study, in patients with bladder cancer who need intravesical therapy. This will allow to optimise the design, assess whether recruitment and interventions are sufficient to allow the trial to progress, and gather preliminary data with the following objectives:

* To determine the safety of T-Control® versus the usual clinical practice in the participating center, by comparing the rate of accidental spillages due to the catheter in patients that require oncological intravesical treatments.
* To determine and compare the usability of T-Control® versus the usual clinical practice in the participating center.

All those patients with bladder cancer who require intravesical treatments with chemotherapy or immunotherapy will be invited to participate and will be interviewed in an initial visit, where the inclusion and exclusion criteria will be checked. The patients will receive information about the study, they will decide whether or not they want to participate, they will sign and deliver the written informed consent and they will be included in the study and randomised into one of the two study interventions. In the subsequent visit, patients will receive the treatment with the alternate catheter. Thus, each patient will receive the intravesical oncological treatment with both catheters assessed in the study.

After the end of each treatment the health professionals who have participated, and after giving their informed consent, will be asked to record all the spillages and leakages occurred during the therapy, whereas at the end of the study they will be asked to measure the usability perceived with both types of catheters

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged ≥18 years.
* Patients with bladder cancer who require intravesical treatments with chemotherapy or immunotherapy.
* Patients requiring recurrent intravesical instillations for their treatment.
* Signed consent agreement.

Exclusion Criteria:

* Patients with difficult catheterisation who require a urologist to perform the catheter insertion.
* Inability to read and understand Portuguese or english.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Rate of accidental spillages | Intravesical therapy procedure (1-2 hours)
  The number of spillages with cytostatics, body fluids or other non-hazardous spillages divided by the number of interventions (intravesical therapy procedures)

SECONDARY OUTCOMES:
General device-usability | Intravesical therapy procedure (1-2 hours)
  The degree of usability perceived by the health professionals involved in the intravesical procedure will be evaluated through the validated USE Questionnaire on more general usability for medical devices.
Specific device-usability | Intravesical therapy procedure (1-2 hours)
  The degree of usability perceived by the health professionals involved in the intravesical procedure will be evaluated through an ad hoc questionnaire on usability during intravesical therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Tiago Santos, Principal Investigator — Champalimaud Clinical Centre

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be available from the Sponsor upon reasonable request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Within one year from the completion of the clinical investigation or three months after its early termination or temporary cessation. When, for scientific reasons, would not possible to submit the clinical research report within one year after completion of the research, it will be submitted as soon as it is available.
Access Criteria: Available from the Sponsor upon reasonable request.